CLINICAL TRIAL: NCT02317471
Title: Immunotherapy of Gastric Cancer With Autologous Tumor Derived Heat Shock Protein gp96
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Cure&Sure Biotech Co., LTD (Industry)
Responsible Party: Principal Investigator, Lin Chen, Director of the general surgery department, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PLAG-CS-Ga-01
Record Dates: First submitted 2014-12-10; First posted 2014-12-16 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Gastric Carcinoma
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gp96 group (Experimental): autologous gp96 vaccination + basal treatment for gastric cancer
  Interventions: Biological: autologous gp96 vaccination; Drug: Oxaliplatin+S-1
- control group (Other): Oxaliplatin+S-1
  Interventions: Drug: Oxaliplatin+S-1

INTERVENTIONS:
Biological: autologous gp96 vaccination — Vaccination of gp96 derived from autologous tumor tissue. Treatment will be started between 3-6 weeks after the surgery.
  gp96 of 25ug in 1mL normal saline s.c. on days 1 of each cycle, up to a maximum of 10 doses (1 cycle= 7 days). 200-400mg cyclophosphamide i.v. 1-3 days before each gp96 infusion.
  Arms: gp96 group
Drug: Oxaliplatin+S-1 — Treatment will be start at the 5th week after the surgery.
  S-1: 40~60mg bid，d1~14 q3W; oxaliplatin:130mg/m2，iv drip for 2h，d1,q3W 6 cycles.
  Other Names: Oxaliplatin(Sanofi-aventis), S-1(Taiho)

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of autologous gp96 treatment of gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Disease characteristics: Histologically confirmed gastric carcinoma: clinical stage III (according to the Japanese gastric cancer classification), must have undergone radical resection
2. Able to read and understand the informed consent document, must sign the informed consent
3. Age: 18 to 75 years old
4. Availability of at least 0.5 g tumor sample
5. ECOG ≤1；life expectancy >=12 weeks, able to comply with study-related procedures
6. Adequate bone marrow function including the absence of lymphopenia (ANC > 1,500/ mm3; Hemoglobin > 10g/dL ; platelet count >100,000/mm3), adequate liver function (serum glutamic oxaloacetic transaminase/ aspartate aminotransferase [AST], alanine amino transferase [ALT] <2.5 times institutional upper limit of normals [IULNs] and bilirubin (total) <1.5 times IULN), and adequate renal function (BUN and creatinine <1.5 times IULNs)
7. Normal heart function
8. NOT participate in ANY other clinical trials within 4 weeks prior to vaccination.

Exclusion Criteria:

1. Unable to get the informed consent
2. Female patients who are pregnant or breastfeeding
3. Progression prior to treatment as determined by the principal investigator
4. Transplant recipient
5. Patients currently diagnosed with Human Immunodeficiency Virus or other active uncontrolled infection
6. Unstable or severe intercurrent medical conditions
7. Patient with allergic constitution
8. Patients with any systemic disease needed to be treated with immunosuppressant or Corticosteroids.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 2 years
Number of participants with adverse events related to gp96 immunotherapy | participants will be followed from the day of the first vaccination to the 30th day after the last vaccination.
  A complete blood count will be requested before the first vaccination, after the second vaccination and after the last vaccination to monitor the side effect of gp96 immunotherapy. And blood chemistries will also be requested at the same time point for the same reason.
  And other adverse events related to gp96 immunotherapy will be recorded according to the NCI-CTCAE 3.0 criteria.

SECONDARY OUTCOMES:
Changes in antigen specific T cells | within 3 days before the first vaccination and within 3 days after the 10th vaccination
  Tumor antigen specific T cells will be determined by IFN-γ Enzyme-linked immunosorbent spot using the autologous tumor cell lysis as the antigen.
Overall survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Lin Chen, MD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China